CLINICAL TRIAL: NCT01620164
Title: Assessment of Three-dimensional Vision Alteration in Parkinson Disease.
Acronym: 3Dparks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1015102; AOL 2010 (Other: CHU de Toulouse)
Record Dates: First submitted 2011-11-07; First posted 2012-06-15 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Parkinson Disease
Keywords: three-dimensional vision; Parkinson
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Parkinsonian patients OFF/ON (Other): 9 patients will be evaluated with psychophysical measurements of 3D perception, in OFF then ON conditions
  Interventions: Other: Psychophysical measurements of 3D perception
- healthy subjects (Other): Healthy subjects will be evaluated with psychophysical measurements of 3D perception, without treatment
  Interventions: Other: Psychophysical measurements of 3D perception
- Parkinsonian patients ON/OFF (Other): 9 patients will be evaluated with psychophysical measurements of 3D perception, in ON and then OFF conditions
  Interventions: Other: Psychophysical measurements of 3D perception

INTERVENTIONS:
Other: Psychophysical measurements of 3D perception — 3D psychophysical performances using a categorization tasks and their underlying mechanisms measured with visual evoked potentials will be assessed in a randomized and comparative study. The order of psychophysical and visual evoked potentials experiments will be randomized between the L Dopa ON and OFF conditions. The randomization will be done by the clinical investigational center. The comparisons will be made between parkinsonian patient and control subjects, and between parkinsonian patients in L Dopa ON and OFF conditions.

SUMMARY:
Parkinson's disease is characterized by motor deficits, improved by dopaminergic intakes. Besides motor symptoms, visual troubles are observed in patients with Parkinson's disease, in particular spatial orientation problems including 3D vision. However, although these visual disturbances are commonly reported by the patients and their family in our clinical experience, they have not been the subject of specific clinical studies yet.

Parkinsonian patients report deficits in 3D vision leading to a loss of visuomotor ability, locomotor functions and to falls. Despite these frequent complaints, little is known about 3D vision in Parkinson's disease. The investigators want in this project to precisely estimate 3D deficits in parkinsonian patients by assessing their psychophysical performances in 3D vision tasks to compare to age matched control subjects' performances.

DETAILED DESCRIPTION:
This is a monocentric and prospective study that will compare Parkinsonian patients versus healthy subjects on the execution of psychophysical tests and Visual Evoked Potentials without and with L Dopa. The comparison will focus on one hand between PD patients and control subjects (matched by age and sex to parkinsonian patients) and on the other hand between parkinsonian patients in ON and OFF drug conditions.

Psychophysical measurements of 3D perception will be performed during this study. This will be done by asking the subjects to indicate with a joystick whether they perceived the stimulus presented on the screen placed in front of them like being 2D or 3D. Two "depth conditions" will be tested; 2D for flat stimuli and 3D for in depth stimuli. Two "3D-cues" conditions will be tested: binocular cues (retinal disparity) and monocular cues (perspective). Their performances will be assessed in both L Dopa ON and OFF conditions randomly determined.

While subjects will be performing the psychophysical tasks, we will record the visual potentials evoked by the presentation of the 2D/3D visual stimuli. Visual Evoked Potentials are obtained by extracting from the EEG the electrical signals temporally locked to the visual stimulations.

3D perception is at the intersection of pure visual perception and navigation; indeed, any movement in a familiar or unfamiliar environment requires an adequate balance between the reality of the three-dimensional environing space and its mental representation. So one of the major roles of the visual system is to convert the two-dimensional retinal images into 3 dimensions. With both binocular (retinal disparity, eye vergence) and monocular (perspective, shading ...) cues, the 3D vision can estimate (1) the distance between objects (2) distance between an object and itself, (3) relief or depth of an object. Altering that perception affects the postural and locomotor functions and thus must worsen motor disorders. So far, no systematic studies have been conducted in parkinsonian patients to quantify their 3D perception. Because of the interaction between 3D perception and motor outcomes, we want, in this project, to estimate the 3D visual deficits, to understand the underlying altered processes, to test the effect of L Dopa on these deficits and to specify the relationship between 3D visual and motor deficits.

3D psychophysical performances using a categorization task and their underlying neuronal mechanisms measured with VEP will be assessed in both Parkinsonian patients and control subjects in a randomized and comparative study.

Parkinsonian patients will be hospitalized for less than 48 hours. Patients randomized in order OFF-ON L Dopa condition will arrive at 8 am. They will perform the first part of the experiment in OFF condition. Later they will receive 150% of their usual treatment dose, perform the experiment and leave the hospital. Patients randomized in order ON-OFF will arrive at 8 am to receive 150% of their usual treatment dose and perform the experiment. The following day, they will perform the experiment weaned from any dopaminergic therapy since midnight in OFF condition. They will leave the hospital after receiving their usual treatment dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease of both sex,
* aged between 50 and 75 with an equivalent corrected vision of minimum 7/10 in both eyes. Patients with vision less than 7/10 in one or both eyes.
* Patients with a normal binocular fusion (Bagolini test).

Control subjects of both sex,

- aged between 50 and 75 with an equivalent corrected vision of minimum 7/10 in both eyes.

Exclusion Criteria:

* Patients with non idiopathic Parkinson's disease.
* Patients with vision less than 7/10.
* Patients with significant tremor during periods of blocking (OFF) or abnormal involuntary movements (dyskinesia) during periods of release (ON).
* Patients with visual hallucinations.
* Patients with impaired cognitive function

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
performance (in percent error) in a 2D/3D categorization task of both parkinsonian patients (OFF treatment) and control subjects. | 12 hours after levodopa intake
  before and after levodopa intake for PD patients and once for healthy volunteers

SECONDARY OUTCOMES:
measure of early visual evoked potentials components latency, recorded in parkinsonian patients, in ON and OFF L Dopa conditions, and in control subjects | 12 hours after levodopa intake
  before and after levodopa intake for PD patients and once for healthy volunteers
assessment of 3D psychophysical performance of parkinsonian patients in both ON and OFF L Dopa conditions | 12 hours after levodopa intake
  before and after levodopa intake for PD patients
search for correlation between the severity of motor impairment of parkinsonian patients and the percentage of error in categorization tasks | 12 hours after levodopa intake
  before and after levodopa intake for PD patients
search for correlation between the severity of motor impairment of parkinsonian patients and the increase of early visual evoked potentials components latency | 12 hours after levodopa intake
  before and after levodopa intake for PD patients

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Ory-Magne, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Hôpital Purpan, Toulouse, France

REFERENCES:
- [Result] Severac Cauquil A, Ory-Magne F, Jardine V, Galitzky M, Rosito M, Brefel-Courbon C, Celebrini S. Parkinson's patients can rely on perspective cues to perceive 3D space. Brain Res. 2017 May 15;1663:161-165. doi: 10.1016/j.brainres.2017.03.017. Epub 2017 Mar 19. PMID 28327351